CLINICAL TRIAL: NCT04695249
Title: Targeting Avoidant Behaviours in Anxiety Disorders Using Individualized 360° Videos: a Multiple Single Case Design
Brief Title: Using 360° Videos in the Treatment of Anxiety Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Clara DELLA LIBERA, Principal Investigator, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-360
Record Dates: First submitted 2020-12-22; First posted 2021-01-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Social Anxiety Disorder; Agoraphobia
Keywords: 360-degree videos; Virtual reality; Exposure therapy; Anxiety disorders
MeSH Terms: conditions — Phobia, Social; Agoraphobia; Anxiety Disorders

STUDY DESIGN:
Masking Description: All assessment pre-post and follow up were realized by an external assessor. The results were blinded to the main psychotherapist (and investigator) until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure intervention (Experimental): Eleven individual sessions.
  Interventions: Behavioral: Exposure intervention using 360 degree videos

INTERVENTIONS:
Behavioral: Exposure intervention using 360 degree videos — The intervention consists of eleven sessions. The first five sessions are dedicated to functional assessment and psychoeducation. The second five sessions are dedicated to exposure in 360-degree videos. The last session is provided for relapse prevention.

SUMMARY:
This study aims to test the feasibility and efficacy of an individualized exposure intervention using 360-degree videos for social anxiety and agoraphobia. A multiple single case design is followed with a pre-post-follow up assessment and multiple baselines. In addition, an experience sampling method is used to explore the role of dysfunctional beliefs and self-efficacy in the efficacy intervention.

DETAILED DESCRIPTION:
There is growing evidence that supports the use of Virtual Reality (VR) to address anxiety disorders such as social anxiety and agoraphobia. The main advantage of VR is to expose participants to their fears in a controlled and safe environment. However, the access to VR remains costly for health professionals who need to pay licenses for the use of a limited number of environments. Therefore, these standardized environments only address the symptoms of standard anxious patients. As a way to provide an accessible tool that can be tailored according to patients' specific difficulties, the proposed approach builds on 360-degree videos as an alternative to VR.

The aim of the present study is to test the feasibility and efficacy of an individualized expo-sure intervention using 360-degree videos. In addition, the role of cognitive processes (i.e., dysfunctional beliefs and self-efficacy) in the exposure efficacy is examined. The intervention includes eleven sessions including five sessions of exposure in 360-degree videos de-signed especially for each patient difficulties.

A multiple single-case design (n=5) is adopted with three types of evaluations: (1) traditional assessment scale of primary/secondary outcomes and aspects related to the therapy, (2) daily ambulatory assessment with a multiple baseline design, (3) experience sampling of cognitive processes about feared situations.

Each video will also be assessed by the participants after exposure sessions.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnostic (DSM 5) of social anxiety or agoraphobia
* High level of avoidance
* French-speaking
* Having a mobile phone which met VR reading criteria

Exclusion Criteria:

* Having a history of psychotic or bipolar disorder
* Having a history of severe brain trauma or epilepsy
* Having a history of respiratory disturbances
* With a concurrent additional psychotherapy
* With acute suicidal ideation
* With a primary diagnosis of depression
* With a non stabilized medication
* Auto medication with alcohol or other substances
* Having migraine or motion sickness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Social anxiety: avoidance | Baseline : up to 4 weeks before intervention
  The French version of the LSAS-SR was used to assess the levels of anxiety and avoidance associated with social situations. The LSAS-SR consists of 24 items describing four types of situations: (1) social interactions, (2) public speaking, (3) eating and drinking in public, (4) being observed. Each item is rated on a 3-point scale according to both the level of fear (0 = "no fear" to 3 = "severe") and the level of avoidance (0 = "never" to 3 = "Usually"). A general total score can be obtained by summing all items and specific score of avoidance and fear as well as scores for specific type of situations can be obtained by summing specific items.
Social anxiety: avoidance | Baseline : up to 3 weeks before intervention
  The French version of the LSAS-SR was used to assess the levels of anxiety and avoidance associated with social situations. The LSAS-SR consists of 24 items describing four types of situations: (1) social interactions, (2) public speaking, (3) eating and drinking in public, (4) being observed. Each item is rated on a 3-point scale according to both the level of fear (0 = "no fear" to 3 = "severe") and the level of avoidance (0 = "never" to 3 = "Usually"). A general total score can be obtained by summing all items and specific score of avoidance and fear as well as scores for specific type of situations can be obtained by summing specific items.
Social anxiety: avoidance | Baseline : up to 2 weeks before intervention
  The French version of the LSAS-SR was used to assess the levels of anxiety and avoidance associated with social situations. The LSAS-SR consists of 24 items describing four types of situations: (1) social interactions, (2) public speaking, (3) eating and drinking in public, (4) being observed. Each item is rated on a 3-point scale according to both the level of fear (0 = "no fear" to 3 = "severe") and the level of avoidance (0 = "never" to 3 = "Usually"). A general total score can be obtained by summing all items and specific score of avoidance and fear as well as scores for specific type of situations can be obtained by summing specific items.
Social anxiety: avoidance | Post intervention : last day of intervention, week 11
  The French version of the LSAS-SR was used to assess the levels of anxiety and avoidance associated with social situations. The LSAS-SR consists of 24 items describing four types of situations: (1) social interactions, (2) public speaking, (3) eating and drinking in public, (4) being observed. Each item is rated on a 3-point scale according to both the level of fear (0 = "no fear" to 3 = "severe") and the level of avoidance (0 = "never" to 3 = "Usually"). A general total score can be obtained by summing all items and specific score of avoidance and fear as well as scores for specific type of situations can be obtained by summing specific items.
Social anxiety: avoidance | Post intervention : 1 week after intervention
  The French version of the LSAS-SR was used to assess the levels of anxiety and avoidance associated with social situations. The LSAS-SR consists of 24 items describing four types of situations: (1) social interactions, (2) public speaking, (3) eating and drinking in public, (4) being observed. Each item is rated on a 3-point scale according to both the level of fear (0 = "no fear" to 3 = "severe") and the level of avoidance (0 = "never" to 3 = "Usually"). A general total score can be obtained by summing all items and specific score of avoidance and fear as well as scores for specific type of situations can be obtained by summing specific items.
Social anxiety: avoidance | Post intervention : 2 week after intervention
  The French version of the LSAS-SR was used to assess the levels of anxiety and avoidance associated with social situations. The LSAS-SR consists of 24 items describing four types of situations: (1) social interactions, (2) public speaking, (3) eating and drinking in public, (4) being observed. Each item is rated on a 3-point scale according to both the level of fear (0 = "no fear" to 3 = "severe") and the level of avoidance (0 = "never" to 3 = "Usually"). A general total score can be obtained by summing all items and specific score of avoidance and fear as well as scores for specific type of situations can be obtained by summing specific items.
Social anxiety: avoidance | Follow up : Three months after intervention
  The French version of the LSAS-SR was used to assess the levels of anxiety and avoidance associated with social situations. The LSAS-SR consists of 24 items describing four types of situations: (1) social interactions, (2) public speaking, (3) eating and drinking in public, (4) being observed. Each item is rated on a 3-point scale according to both the level of fear (0 = "no fear" to 3 = "severe") and the level of avoidance (0 = "never" to 3 = "Usually"). A general total score can be obtained by summing all items and specific score of avoidance and fear as well as scores for specific type of situations can be obtained by summing specific items.
Social anxiety: avoidance | Follow up : 3 months and 1 week after intervention
  The French version of the LSAS-SR was used to assess the levels of anxiety and avoidance associated with social situations. The LSAS-SR consists of 24 items describing four types of situations: (1) social interactions, (2) public speaking, (3) eating and drinking in public, (4) being observed. Each item is rated on a 3-point scale according to both the level of fear (0 = "no fear" to 3 = "severe") and the level of avoidance (0 = "never" to 3 = "Usually"). A general total score can be obtained by summing all items and specific score of avoidance and fear as well as scores for specific type of situations can be obtained by summing specific items.
Social anxiety: avoidance | Follow up : 3 months and 2 weeks after intervention
  The French version of the LSAS-SR was used to assess the levels of anxiety and avoidance associated with social situations. The LSAS-SR consists of 24 items describing four types of situations: (1) social interactions, (2) public speaking, (3) eating and drinking in public, (4) being observed. Each item is rated on a 3-point scale according to both the level of fear (0 = "no fear" to 3 = "severe") and the level of avoidance (0 = "never" to 3 = "Usually"). A general total score can be obtained by summing all items and specific score of avoidance and fear as well as scores for specific type of situations can be obtained by summing specific items.
Social anxiety: severity | Baseline : up to 4 weeks before intervention
  The French version of the SIAS was used to assess social anxiety severity. The SIAS consists of 20 self-statements describing one's reaction to situations that involve social interaction. Each item is rated on a 4-point Likert scale ranging from 0 = "not at all characteristic or true of me" to 4 "extremely characteristic or true of me". The SIAS is scored by summing the ratings. Total score ranges from 0 to 80, with higher scores representing higher levels of social interaction anxiety.
Social anxiety: severity | Baseline : up to 3 weeks before intervention
  The French version of the SIAS was used to assess social anxiety severity. The SIAS consists of 20 self-statements describing one's reaction to situations that involve social interaction. Each item is rated on a 4-point Likert scale ranging from 0 = "not at all characteristic or true of me" to 4 "extremely characteristic or true of me". The SIAS is scored by summing the ratings. Total score ranges from 0 to 80, with higher scores representing higher levels of social interaction anxiety.
Social anxiety: severity | Baseline : up to 2 weeks before intervention
  The French version of the SIAS was used to assess social anxiety severity. The SIAS consists of 20 self-statements describing one's reaction to situations that involve social interaction. Each item is rated on a 4-point Likert scale ranging from 0 = "not at all characteristic or true of me" to 4 "extremely characteristic or true of me". The SIAS is scored by summing the ratings. Total score ranges from 0 to 80, with higher scores representing higher levels of social interaction anxiety.
Social anxiety: severity | Post intervention : last day of intervention, week 11
  The French version of the SIAS was used to assess social anxiety severity. The SIAS consists of 20 self-statements describing one's reaction to situations that involve social interaction. Each item is rated on a 4-point Likert scale ranging from 0 = "not at all characteristic or true of me" to 4 "extremely characteristic or true of me". The SIAS is scored by summing the ratings. Total score ranges from 0 to 80, with higher scores representing higher levels of social interaction anxiety.
Social anxiety: severity | Post intervention : 1 week after intervention
  The French version of the SIAS was used to assess social anxiety severity. The SIAS consists of 20 self-statements describing one's reaction to situations that involve social interaction. Each item is rated on a 4-point Likert scale ranging from 0 = "not at all characteristic or true of me" to 4 "extremely characteristic or true of me". The SIAS is scored by summing the ratings. Total score ranges from 0 to 80, with higher scores representing higher levels of social interaction anxiety.
Social anxiety: severity | Post intervention : 2 week after intervention
  The French version of the SIAS was used to assess social anxiety severity. The SIAS consists of 20 self-statements describing one's reaction to situations that involve social interaction. Each item is rated on a 4-point Likert scale ranging from 0 = "not at all characteristic or true of me" to 4 "extremely characteristic or true of me". The SIAS is scored by summing the ratings. Total score ranges from 0 to 80, with higher scores representing higher levels of social interaction anxiety.
Social anxiety: severity | Follow up : 3 months after intervention
  The French version of the SIAS was used to assess social anxiety severity. The SIAS consists of 20 self-statements describing one's reaction to situations that involve social interaction. Each item is rated on a 4-point Likert scale ranging from 0 = "not at all characteristic or true of me" to 4 "extremely characteristic or true of me". The SIAS is scored by summing the ratings. Total score ranges from 0 to 80, with higher scores representing higher levels of social interaction anxiety.
Social anxiety: severity | Follow up : 3 months and 1 week after intervention
  The French version of the SIAS was used to assess social anxiety severity. The SIAS consists of 20 self-statements describing one's reaction to situations that involve social interaction. Each item is rated on a 4-point Likert scale ranging from 0 = "not at all characteristic or true of me" to 4 "extremely characteristic or true of me". The SIAS is scored by summing the ratings. Total score ranges from 0 to 80, with higher scores representing higher levels of social interaction anxiety.
Social anxiety: severity | Follow up : 3 months and 2 week after intervention
  The French version of the SIAS was used to assess social anxiety severity. The SIAS consists of 20 self-statements describing one's reaction to situations that involve social interaction. Each item is rated on a 4-point Likert scale ranging from 0 = "not at all characteristic or true of me" to 4 "extremely characteristic or true of me". The SIAS is scored by summing the ratings. Total score ranges from 0 to 80, with higher scores representing higher levels of social interaction anxiety.
Agoraphobia: avoidance | Baseline : up to 4 weeks before intervention
  The French version of the MIA was used to assess the levels of agoraphobic avoidance. The MIA consists of 25 items describing agoraphobic situations. Each item is rated according to the level of avoidance on a 5-point Likert scale ranging from 1 = "never avoid" to 5 = "always avoid", both when the participants are accompanied or alone. One final question concerns the number of panic attacks during the last week. The MIA provides a score for situations alone or accompanied by summing the ratings. Higher scores indicate higher levels of avoidance.
Agoraphobia: avoidance | Baseline : up to 3 weeks before intervention
  The French version of the MIA was used to assess the levels of agoraphobic avoidance. The MIA consists of 25 items describing agoraphobic situations. Each item is rated according to the level of avoidance on a 5-point Likert scale ranging from 1 = "never avoid" to 5 = "always avoid", both when the participants are accompanied or alone. One final question concerns the number of panic attacks during the last week. The MIA provides a score for situations alone or accompanied by summing the ratings. Higher scores indicate higher levels of avoidance.
Agoraphobia: avoidance | Baseline : up to 2 weeks before intervention
  The French version of the MIA was used to assess the levels of agoraphobic avoidance. The MIA consists of 25 items describing agoraphobic situations. Each item is rated according to the level of avoidance on a 5-point Likert scale ranging from 1 = "never avoid" to 5 = "always avoid", both when the participants are accompanied or alone. One final question concerns the number of panic attacks during the last week. The MIA provides a score for situations alone or accompanied by summing the ratings. Higher scores indicate higher levels of avoidance.
Agoraphobia: avoidance | Post intervention : last day of intervention, week 11
  The French version of the MIA was used to assess the levels of agoraphobic avoidance. The MIA consists of 25 items describing agoraphobic situations. Each item is rated according to the level of avoidance on a 5-point Likert scale ranging from 1 = "never avoid" to 5 = "always avoid", both when the participants are accompanied or alone. One final question concerns the number of panic attacks during the last week. The MIA provides a score for situations alone or accompanied by summing the ratings. Higher scores indicate higher levels of avoidance.
Agoraphobia: avoidance | Post intervention : 1 week after intervention
  The French version of the MIA was used to assess the levels of agoraphobic avoidance. The MIA consists of 25 items describing agoraphobic situations. Each item is rated according to the level of avoidance on a 5-point Likert scale ranging from 1 = "never avoid" to 5 = "always avoid", both when the participants are accompanied or alone. One final question concerns the number of panic attacks during the last week. The MIA provides a score for situations alone or accompanied by summing the ratings. Higher scores indicate higher levels of avoidance.
Agoraphobia: avoidance | Post intervention : 2 week after intervention
  The French version of the MIA was used to assess the levels of agoraphobic avoidance. The MIA consists of 25 items describing agoraphobic situations. Each item is rated according to the level of avoidance on a 5-point Likert scale ranging from 1 = "never avoid" to 5 = "always avoid", both when the participants are accompanied or alone. One final question concerns the number of panic attacks during the last week. The MIA provides a score for situations alone or accompanied by summing the ratings. Higher scores indicate higher levels of avoidance.
Agoraphobia: avoidance | Follow up : 3 months after intervention
  The French version of the MIA was used to assess the levels of agoraphobic avoidance. The MIA consists of 25 items describing agoraphobic situations. Each item is rated according to the level of avoidance on a 5-point Likert scale ranging from 1 = "never avoid" to 5 = "always avoid", both when the participants are accompanied or alone. One final question concerns the number of panic attacks during the last week. The MIA provides a score for situations alone or accompanied by summing the ratings. Higher scores indicate higher levels of avoidance.
Agoraphobia: avoidance | Follow up : 3 months and 1 week after intervention
  The French version of the MIA was used to assess the levels of agoraphobic avoidance. The MIA consists of 25 items describing agoraphobic situations. Each item is rated according to the level of avoidance on a 5-point Likert scale ranging from 1 = "never avoid" to 5 = "always avoid", both when the participants are accompanied or alone. One final question concerns the number of panic attacks during the last week. The MIA provides a score for situations alone or accompanied by summing the ratings. Higher scores indicate higher levels of avoidance.
Agoraphobia: avoidance | Follow up : 3 months and 2 weeks after intervention
  The French version of the MIA was used to assess the levels of agoraphobic avoidance. The MIA consists of 25 items describing agoraphobic situations. Each item is rated according to the level of avoidance on a 5-point Likert scale ranging from 1 = "never avoid" to 5 = "always avoid", both when the participants are accompanied or alone. One final question concerns the number of panic attacks during the last week. The MIA provides a score for situations alone or accompanied by summing the ratings. Higher scores indicate higher levels of avoidance.
Agoraphobia: Severity | Baseline : up to 4 weeks before intervention
  The French version of the Panic and Agoraphobia Scale consists of 13 items divided in five subscales: (1) panic attacks, (2) agoraphobia, (3) anticipatory anxiety, (4) interference with family/hobbies/working and (5) worries about health. Each item is rated on a specific 5-point scale, with higher scores indicating higher severity. The PAS is scored by summing the subscales and all items with a total score ranging from 13 to 52.
Agoraphobia: Severity | Baseline : up to 3 weeks before intervention
  The French version of the Panic and Agoraphobia Scale consists of 13 items divided in five subscales: (1) panic attacks, (2) agoraphobia, (3) anticipatory anxiety, (4) interference with family/hobbies/working and (5) worries about health. Each item is rated on a specific 5-point scale, with higher scores indicating higher severity. The PAS is scored by summing the subscales and all items with a total score ranging from 13 to 52.
Agoraphobia: Severity | Baseline : up to 2 weeks before intervention
  The French version of the Panic and Agoraphobia Scale consists of 13 items divided in five subscales: (1) panic attacks, (2) agoraphobia, (3) anticipatory anxiety, (4) interference with family/hobbies/working and (5) worries about health. Each item is rated on a specific 5-point scale, with higher scores indicating higher severity. The PAS is scored by summing the subscales and all items with a total score ranging from 13 to 52.
Agoraphobia: Severity | Post intervention : last day of intervention, week 11
  The French version of the Panic and Agoraphobia Scale consists of 13 items divided in five subscales: (1) panic attacks, (2) agoraphobia, (3) anticipatory anxiety, (4) interference with family/hobbies/working and (5) worries about health. Each item is rated on a specific 5-point scale, with higher scores indicating higher severity. The PAS is scored by summing the subscales and all items with a total score ranging from 13 to 52.
Agoraphobia: Severity | Post intervention : 1 week after intervention
  The French version of the Panic and Agoraphobia Scale consists of 13 items divided in five subscales: (1) panic attacks, (2) agoraphobia, (3) anticipatory anxiety, (4) interference with family/hobbies/working and (5) worries about health. Each item is rated on a specific 5-point scale, with higher scores indicating higher severity. The PAS is scored by summing the subscales and all items with a total score ranging from 13 to 52.
Agoraphobia: Severity | Post intervention : 2 week after intervention
  The French version of the Panic and Agoraphobia Scale consists of 13 items divided in five subscales: (1) panic attacks, (2) agoraphobia, (3) anticipatory anxiety, (4) interference with family/hobbies/working and (5) worries about health. Each item is rated on a specific 5-point scale, with higher scores indicating higher severity. The PAS is scored by summing the subscales and all items with a total score ranging from 13 to 52.
Agoraphobia: Severity | Follow up : 3 months after intervention
  The French version of the Panic and Agoraphobia Scale consists of 13 items divided in five subscales: (1) panic attacks, (2) agoraphobia, (3) anticipatory anxiety, (4) interference with family/hobbies/working and (5) worries about health. Each item is rated on a specific 5-point scale, with higher scores indicating higher severity. The PAS is scored by summing the subscales and all items with a total score ranging from 13 to 52.
Agoraphobia: Severity | Follow up : 3 months and 1 week after intervention
  The French version of the Panic and Agoraphobia Scale consists of 13 items divided in five subscales: (1) panic attacks, (2) agoraphobia, (3) anticipatory anxiety, (4) interference with family/hobbies/working and (5) worries about health. Each item is rated on a specific 5-point scale, with higher scores indicating higher severity. The PAS is scored by summing the subscales and all items with a total score ranging from 13 to 52.
Agoraphobia: Severity | Follow up : 3 months and 2 weeks after intervention
  The French version of the Panic and Agoraphobia Scale consists of 13 items divided in five subscales: (1) panic attacks, (2) agoraphobia, (3) anticipatory anxiety, (4) interference with family/hobbies/working and (5) worries about health. Each item is rated on a specific 5-point scale, with higher scores indicating higher severity. The PAS is scored by summing the subscales and all items with a total score ranging from 13 to 52.
Multiple measures for change in levels of anxiety | Baseline : 1x/day (up to 3 week before the intervention)
  A questionnaire comprising four questions regarding the daily rate of avoidant behaviours, approach behaviours, level of anxiety and the severity of anxiety consequences. The questionnaire was sent every day to the participant via a mobile app. Higher scores indicate higher levels of avoidance, approach, anxiety and severity of anxiety consequences.
Multiple measures for change in levels of anxiety | Intervention : 1x/day (11weeks)
  A questionnaire comprising four questions regarding the daily rate of avoidant behaviours, approach behaviours, level of anxiety and the severity of anxiety consequences. The questionnaire was sent every day to the participant via a mobile app. Higher scores indicate higher levels of avoidance, approach, anxiety and severity of anxiety consequences.
Multiple measures for change in levels of anxiety | Post-intervention : 1x/day (3 weeks)
  A questionnaire comprising four questions regarding the daily rate of avoidant behaviours, approach behaviours, level of anxiety and the severity of anxiety consequences. The questionnaire was sent every day to the participant via a mobile app. Higher scores indicate higher levels of avoidance, approach, anxiety and severity of anxiety consequences.

SECONDARY OUTCOMES:
Depression Anxiety and Stress | Baseline : up to three weeks before intervention
  The DASS consists of 21 items assessing (1) depression, (2) anxiety and (3) stress with self-statement. With reference to the last week, all items are rated on a 4-point Likert scale ranging from 0 = "Did not apply to me at all" to 3 "Applied to me very much or most of the time". Scores for each subscale are obtained by summing the scores of relevant items. Higher scores indicate higher level of depression, anxiety and stress.
Depression Anxiety and Stress | Post intervention : 1 weeks after intervention
  The DASS consists of 21 items assessing (1) depression, (2) anxiety and (3) stress with self-statement. With reference to the last week, all items are rated on a 4-point Likert scale ranging from 0 = "Did not apply to me at all" to 3 "Applied to me very much or most of the time". Scores for each subscale are obtained by summing the scores of relevant items. Higher scores indicate higher level of depression, anxiety and stress.
Depression Anxiety and Stress | Follow up : 3 months after intervention
  The DASS consists of 21 items assessing (1) depression, (2) anxiety and (3) stress with self-statement. With reference to the last week, all items are rated on a 4-point Likert scale ranging from 0 = "Did not apply to me at all" to 3 "Applied to me very much or most of the time". Scores for each subscale are obtained by summing the scores of relevant items. Higher scores indicate higher level of depression, anxiety and stress.
Self-efficacy toward managing the situation, the occurrence of the feared outcome and the fear itself | Baseline : up to three weeks before intervention
  A non-validated French version of the ACQ-R was used to assess the participants' perception of control over anxiety and anxiety-related situations (i.e. similar to self-efficacy). The ACQ-R is a 15-items scale assessing the perceived control of (1) emotion (5 items; e.g., "I am able to control my level of anxiety"), (2) threats (6 items; e.g., "There is little I can do to change frightening events") and (3) stress (4 items; e.g., "When I a put under stress, I am likely to lose control").
Self-efficacy toward managing the situation, the occurrence of the feared outcome and the fear itself | Post intervention : 1 weeks after intervention
  A non-validated French version of the ACQ-R was used to assess the participants' perception of control over anxiety and anxiety-related situations (i.e. similar to self-efficacy). The ACQ-R is a 15-items scale assessing the perceived control of (1) emotion (5 items; e.g., "I am able to control my level of anxiety"), (2) threats (6 items; e.g., "There is little I can do to change frightening events") and (3) stress (4 items; e.g., "When I a put under stress, I am likely to lose control").
Self-efficacy toward managing the situation, the occurrence of the feared outcome and the fear itself | Follow up : 3 months after intervention
  A non-validated French version of the ACQ-R was used to assess the participants' perception of control over anxiety and anxiety-related situations (i.e. similar to self-efficacy). The ACQ-R is a 15-items scale assessing the perceived control of (1) emotion (5 items; e.g., "I am able to control my level of anxiety"), (2) threats (6 items; e.g., "There is little I can do to change frightening events") and (3) stress (4 items; e.g., "When I a put under stress, I am likely to lose control").
Dysfunctional beliefs | Baseline : up to three weeks before intervention
  A non-validated French version of the AABS-2 was used to assess dysfunctional beliefs known to be aetiologically related to anxiety. The AABS-2 consists of 33 beliefs concerning (1) Exposure to judgement, (2) Body vigilance, (3) Thought manifestations and (4) Anxiety. Items are rated on a 7-point Likert scale ranging from 0 to 100 with anchor points at 20, 40, 50, 60, 80%. The four specific scores and one general score are obtained by adding the relevant items. Higher scores indicate greater adherence in beliefs associated with anxiety.
Dysfunctional beliefs | Post intervention : 1 weeks after intervention
  A non-validated French version of the AABS-2 was used to assess dysfunctional beliefs known to be aetiologically related to anxiety. The AABS-2 consists of 33 beliefs concerning (1) Exposure to judgement, (2) Body vigilance, (3) Thought manifestations and (4) Anxiety. Items are rated on a 7-point Likert scale ranging from 0 to 100 with anchor points at 20, 40, 50, 60, 80%. The four specific scores and one general score are obtained by adding the relevant items. Higher scores indicate greater adherence in beliefs associated with anxiety.
Dysfunctional beliefs | Follow up : 3 months after intervention
  A non-validated French version of the AABS-2 was used to assess dysfunctional beliefs known to be aetiologically related to anxiety. The AABS-2 consists of 33 beliefs concerning (1) Exposure to judgement, (2) Body vigilance, (3) Thought manifestations and (4) Anxiety. Items are rated on a 7-point Likert scale ranging from 0 to 100 with anchor points at 20, 40, 50, 60, 80%. The four specific scores and one general score are obtained by adding the relevant items. Higher scores indicate greater adherence in beliefs associated with anxiety.
Therapy outcome | Baseline : up to three weeks before intervention
  The French version of the outcome Questionnaire was used to assess clinical changes in participants. The MI-45 consists of 45 items that assess (1) intrapsychic symptoms of distress (i.e., 25 items, symptoms of depression and anxiety) (2) interpersonal relationship, (i.e., 11 items, satisfaction and difficulties during social interactions) and (3) social roles performance (i.e., 9 items, level of dissatisfaction, conflict, distress and incompetence related to employment, family and hobbies). All items are rated on a 5-point Likert scale ranging from 0 = Never to 4 = Almost Always. The total score ranging from 0 to 80 and the three specific scores can be obtained by adding the relevant items. In addition, the scale possesses a clinical threshold of 63 and a "reliable clinical change" starting from a 17-points gain or loss.
Therapy outcome | Post intervention : 1 weeks after intervention
  The French version of the outcome Questionnaire was used to assess clinical changes in participants. The MI-45 consists of 45 items that assess (1) intrapsychic symptoms of distress (i.e., 25 items, symptoms of depression and anxiety) (2) interpersonal relationship, (i.e., 11 items, satisfaction and difficulties during social interactions) and (3) social roles performance (i.e., 9 items, level of dissatisfaction, conflict, distress and incompetence related to employment, family and hobbies). All items are rated on a 5-point Likert scale ranging from 0 = Never to 4 = Almost Always. The total score ranging from 0 to 80 and the three specific scores can be obtained by adding the relevant items. In addition, the scale possesses a clinical threshold of 63 and a "reliable clinical change" starting from a 17-points gain or loss.
Therapy outcome | Follow up : 3 months after intervention
  The French version of the outcome Questionnaire was used to assess clinical changes in participants. The MI-45 consists of 45 items that assess (1) intrapsychic symptoms of distress (i.e., 25 items, symptoms of depression and anxiety) (2) interpersonal relationship, (i.e., 11 items, satisfaction and difficulties during social interactions) and (3) social roles performance (i.e., 9 items, level of dissatisfaction, conflict, distress and incompetence related to employment, family and hobbies). All items are rated on a 5-point Likert scale ranging from 0 = Never to 4 = Almost Always. The total score ranging from 0 to 80 and the three specific scores can be obtained by adding the relevant items. In addition, the scale possesses a clinical threshold of 63 and a "reliable clinical change" starting from a 17-points gain or loss.
Multiple measures of transfer and control variables | Baseline : 1x/day (up to three weeks before intervention )
  A questionnaire comprising 13 questions regarding the daily rate of positive and negative affects, the specific objective of the participant and control. The questionnaire was sent every day to the participant via a mobile app.
Multiple measures of transfer and control variables | Intervention : 1x/day (11weeks)
  A questionnaire comprising 13 questions regarding the daily rate of positive and negative affects, the specific objective of the participant and control. The questionnaire was sent every day to the participant via a mobile app.
Multiple measures of transfer and control variables | Post-intervention : 1x/day (3 weeks)
  A questionnaire comprising 13 questions regarding the daily rate of positive and negative affects, the specific objective of the participant and control. The questionnaire was sent every day to the participant via a mobile app.
Experience sampling method | Baseline : up to 5x/day (up to 21 days)
  Questionaire including 8 to 11 questions (3 conditioned) regarding the nature, response and appraisal of anxious situations. Participants were asked to reply to the questionnaire on a mobile app when facing feared situations.
Experience sampling method | Intervention : up to 5x/day (11 weeks)
  Questionaire including 8 to 11 questions (3 conditioned) regarding the nature, response and appraisal of anxious situations. Participants were asked to reply to the questionnaire on a mobile app when facing feared situations.
Experience sampling method | Post-intervention : spontaneous responses during 2 weeks after intervention
  Questionaire including 8 to 11 questions (3 conditioned) regarding the nature, response and appraisal of anxious situations. Participants were asked to reply to the questionnaire on a mobile app when facing feared situations.

OTHER OUTCOMES:
Credibility and expectancy of treatment | Baseline : up to three weeks before intervention
  The French version of the Credibility and Expectancies Questionnaire (CEQ) was used at pre and post-assessment. The CEQ consists of 6 items that assess (1) the therapy credibility (i.e., the extent to which the treatment makes sense, is believable, convincing and logical) and (2) expectancies towards the therapy (i.e., improvements expected through the intervention). Higher scores indicate higher credibility and positive expectancies towards the treatment. Higher scores indicate higher credibility and positive expectancies towards the treatment.
Credibility and expectancy of treatment | Post intervention : 1 weeks after intervention
  The French version of the Credibility and Expectancies Questionnaire (CEQ) was used at pre and post-assessment. The CEQ consists of 6 items that assess (1) the therapy credibility (i.e., the extent to which the treatment makes sense, is believable, convincing and logical) and (2) expectancies towards the therapy (i.e., improvements expected through the intervention). Higher scores indicate higher credibility and positive expectancies towards the treatment. Higher scores indicate higher credibility and positive expectancies towards the treatment.
Client Satisfaction towards the treatment | Post intervention : 1 weeks after intervention
  The Client Satisfaction Questionnaire (CSQ) consists of 8-items that assess client satisfaction with treatment. Higher scores indicate greater client satisfaction and therapeutic alliance. Higher scores indicate higher levels of satisfaction towards the treatment.
Helping Alliance | Post intervention : 1 weeks after intervention
  The Helping Alliance Questionnaire (HAQ) consist of 8-items that assess the quality of the therapeutic alliance. Higher scores indicate greater therapeutic alliance. Higher scores indicate higher levels of therapeutic alliance.
Therapy-related evaluation | Intervention phase : 1x/week (11 week)
  A questionnaire including three questions about the therapeutic alliance, therapy credibility, and therapy satisfaction. The participant received the questionnaire once a week on a mobile ap. Higher scores indicate higher satisfaction, credibility and therapeutic alliance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No
Data and analyses will be available from an online repository or from the principal investigator